CLINICAL TRIAL: NCT03314844
Title: Plasma Glucagon-like Peptide-1 Levels Predict In-hospital Complications in ST-segment Elevation Myocardial Infarction
Brief Title: Plasma Glucagon-like Peptide-1 Levels and In-hospital Complications in ST-segment Elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Jing Wei, doctor, Chinese PLA General Hospital
Other Study IDs: GLP1-IHC
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Glucagon-like Peptide-1; Bleeding; Complications
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Glucagon-like peptide-1 (GLP-1), produced mainly in enteroendocrine cells, participates in energy homeostasis and glucose metabolism by regulating islet hormone secretion, gastrointestinal motility, and food intake, making GLP-1 agonist a treatment for diabetes and obesity. Pre-clinical and clinical studies have demonstrated that GLP-1 also has cardio-protection effects. GLP-1 agonists is able to improve markers of cardiac function, reduce myocardial infarct size and post-myocardial infarction remodeling in experimental myocardial infarction. And GLP-1 infusion improved left ventricular function and increases myocardial salvage in patients with acute myocardial infarction (AMI). The investigators' previous study found that GLP-1 analogues attenuated ischemia-reperfusion induced apoptosis of stem- and myocardial microvascular endothelial cells, and liraglutide (a GLP-1 analog) usage during hospital stay can prevent no-reflow and improve heart function in AMI. Therefore, the investigators carried out a cohort study to evaluate the association between plasma GLP-1 and in-hospital complications in patients with ST-segment elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of STEMI and needed PCI

Exclusion Criteria:

* patients with cancer patients who used DPP4 inhibitor patients who used GLP1 analogue

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PLA general hospital (PLAGH) is a large national tertiary-care center in the Beijing, China. The investigators enrolled all patients consecutively hospitalized in PLAGH, with a diagnosis of STEMI and needed PCI
Sampling Method: Non-Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
in-hospital complications | Time Frame: up to 2 week after PCI (until discharge)
  defined as acute heart failure, atrial fibrillation, chest pain or re-acute myocardial infarction, complete atrioventricular block, cerebrovascular disease, ventricular fibrillation or ventricular tachycardia

SECONDARY OUTCOMES:
in-hospital major adverse cardiac or cerebrovascular events | Time Frame: up to 2 week after PCI (until discharge)]
  the composite of death, nonfatal MI, or stroke
in-hospital major bleeding | Time Frame: up to 2 week after PCI (until discharge)
  defined as absolute hemoglobin drop (baseline to nadir)≥4g/dl, intracranial hemorrhage, retroperitoneal hemorrhage, use of red blood cell transfusion in patients with a baseline hemoglobin ≥9.0 g/dl, and use of red blood cell transfusion among patients with a baseline hemoglobin <9.0 g/dl and a witnessed bleeding event